CLINICAL TRIAL: NCT04809337
Title: Comparison of the Effects of Therapeutic Exercises and Stabilization Exercises After Manual Therapy in Patients With Non-Specific Chronic Neck Pain
Brief Title: Therapeutic Exercises and Stabilization Exercises Given After Manual Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Emine Atıcı, Principal Investigator, Okan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 005
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Patients With Non-Specific Chronic Neck Pain
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stabilization Exercise Group (Experimental)
  Interventions: Other: Exercise
- Therapeutic Exercise Group (Experimental)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — After manuel therapy, the patients were allocated into two groups as Stabilization Exercise Group and Therapeutic Exercise Group randomly.

SUMMARY:
The study was conducted to determine and compare the effects of the therapeutic exercises and stabilization exercises given to the patient after the manual therapy session on pain, neck range of motion, daily living activities and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65,
* having neck pain for 3 months or longer,
* was diagnosed with chronic neck pain by a specialist.

Exclusion Criteria:

* People with neurological diseases,
* who had previous surgery in the cervical region,
* who had medulla spinalis tumors,
* vascular pathologies,
* fractures,
* osteoporosis,
* rheumatoid arthritis problems were not included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 1 minute
  The Visual Analog Scale (VAS) was developed to transform values which cannot be measured numerically to a numerical form. The patient is instructed to mark the severity of pain on a line marked at one end as 0=no pain to 10=intolerable pain, thereby providing the level of pain in a numerical form
Range of motion | 10 minute
  Devices to measure range of motion in the joints of the body include the Goniometer and Inclinometer which use a stationary arm, protractor, fulcrum, and movement arm to measure angle from axis of the joint. We measured neck flexio, extantion and rotation

SECONDARY OUTCOMES:
Lateral Scapular Shift Test | 5 minute
  This test involves measuring the distance from the inferior angle of the scapula to the nearest vertebral spinous process using a tape measure or goniometer in three positions: shoulder in neutral, shoulder at 40-45 degrees of coronal plane abduction with hands resting on hips, and the shoulder at 90 degrees abduction with the arms in full internal rotation
Neck Disability Index | 3 minutes
  The Neck Disability Index (NDI) is a self-report questionnaire used to determine how neck pain affects a patient's daily life and to assess the self-rated disability of patients with neck pain
Bournemouth Neck Pain Questionnaire | 5 minutes
  Neck Bournemouth Questionnaire (NBQ) was created by Bolton and Humphreys due to the necessity of an evaluation measure to various health domains, such as pain, function, incapacity and psychological and social aspects of patients with neck pathologies. This tool is easily applied, reproducible and responsive to clinical alterations, which makes it adequate to be used for scientific research and clinical practice to monitor the pathology progression and to assist treatment planning.

CONTACTS AND LOCATIONS:
Locations (1):
- Emine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided